CLINICAL TRIAL: NCT04218734
Title: A Multicenter, Randomized, Double-blind, Parallel Controlled Phase III Clinical Trial of DBRP108 in Combination With Metformin Hydrochloride in the Treatment of Type 2 Diabetes Mellitus
Brief Title: A Study of DBPR108 and Metformin Hydrochloride Combination Therapy in Patients With T2DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPC/DBPR108201903/PRO-III-2
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DBPR108; Dipeptidyl peptidase-4 (DPP4) inhibitors; metformin hydrochloride
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — DBPR108; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin hydrochloride+DBPR108 (Experimental): metformin hydrochloride 500 mg+DBPR108 100 mg
  Interventions: Drug: DBPR108; Drug: metformin hydrochloride
- metformin hydrochloride+placepo (Placebo Comparator): metformin hydrochloride 500 mg+placebo 100 mg
  Interventions: Drug: metformin hydrochloride; Drug: placepo

INTERVENTIONS:
Drug: DBPR108 — DBPR108: 100 mg, once daily for 24 weeks.
  Arms: metformin hydrochloride+DBPR108
Drug: metformin hydrochloride — metformin hydrochloride: 500 mg, 1-3 times daily for 24 weeks.
Drug: placepo — placebo:100 mg, once daily for 24 weeks.
  Arms: metformin hydrochloride+placepo

SUMMARY:
This study aims to evaluate the efficacy and safety of DBPR108 tablets in combination with metformin hydrochloride in the treatment of type 2 diabetes mellitus. A total of 210 subjects will be randomly assigned in a ratio of 2:1 to receive metformin hydrochloride plus DBPR108 or metformin hydrochloride plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes according to World Health Organization (1999) diabetes diagnosis standard;
* Age 18-75 years, men and women;
* BMI 19-35 kg/m2;
* HbA1c 7.0%-9.5%;
* Before screening, a stable Metformin dose（≥1000mg/day）should be maintained for at least 8 weeks.
* Signed informed consent from the patient;
* Agree to use contraceptive measures from the date of signing the informed consent to 1 month after the end of the last medication.

Exclusion Criteria:

* FPG > 13.9 mmol/L;
* Insulin treatment required in the investigator's opinion;
* Administration of antidiabetic drugs (except for metformin) including insulin, rosiglitazone, pioglitazone, DPP-4 inhibitor, Glucagon like peptide-1 (GLP-1) receptor agonist for 8 weeks before screening;
* Acute complications of diabetes (including diabetic ketosis and ketoacidosis, hyperosmotic nonketotic diabetic coma, lactic acidosis and hypoglycemia coma);
* Severe hypoglycemia;
* Serious diabetic complications (such as diabetic foot, etc.);
* History of acute or chronic pancreatitis, or related diseases that are most common cause of acute pancreatitis (such as recurrent cholelithiasis, etc.);
* History of being allergic to DPP-4 inhibitors;
* Untreated hyperthyroidism and other diseases which may cause secondary hyperglycemia;
* Previous treatment with glucocorticoids (except for external use and inhalation) within 4 weeks before screening or may be used for more than 14 consecutive days during the study;
* Inflammatory bowel disease, partial intestinal obstruction or chronic bowel disease related to obvious digestive and absorption disorders;
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 3*upper limit of normal (ULN), or total bilirubin > 1.5ULN;
* Abnormal renal function;
* White blood cells (WBC) < 3.0109/l, neutrophil count of peripheral blood < 1.5109/l, hemoglobin < 100g / L, triglyceride > 5.7 mmol/l;
* HBsAg, HBeAg or HBcAb positive, or any one of hepatitis C antibody, anti-HIV antibody and nonspecific antibody of Treponema pallidum positive;
* Pregnant or lactating women;
* History of alcohol or drug abuse;
* Participation in other clinical trials or administration of any other investigational drugs or devices within 3 months before screening;
* Significant unstable diseases;
* Any condition that in the investigator's opinion might render the patient unable to participate the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (%) from baseline to week 24 | baseline, 24 weeks
  The change of HbA1c from baseline to 24 weeks compared with metformin hydrochloride + placebo

SECONDARY OUTCOMES:
Percentage of HbA1c ≤ 6.5% | 24 weeks
  Proportion of patients achieving HbA1c ≤ 6.5% at week 24
Percentage of HbA1c ≤ 7% | 24 weeks
  Proportion of patients achieving HbA1c ≤ 7% at week 24
Change in HbA1c (%) from baseline to week 12 | baseline, 12 weeks
  The change of HbA1c from baseline to 12 weeks compared with metformin hydrochloride + placebo
Change in fasting plasma glucose (FPG) from baseline to week 12 and week 24 | Baseline, 12 weeks and 24 weeks
  The change in FPG from baseline to week 12 and week 24 compared with metformin hydrochloride + placebo
Change in 2h-postprandial plasma glucose (2h-PPG) from baseline to week 12 and week 24 | Baseline, 12 weeks and 24 weeks
  The change in 2h-PPG from baseline to week 12 and week 24 compared with metformin hydrochloride + placebo
Change in body weight from baseline to week 12 and week 24 | Baseline, 12 weeks and 24 weeks
  The change in body weight from baseline to week 12 and week 24 compared with metformin hydrochloride +placebo

CONTACTS AND LOCATIONS:
Overall Officials: Kun Lou, Study Director — Department of medicine, CSPC clinical development division
Locations (1):
- Peking Union Medical College Hospital, Beijing, China